CLINICAL TRIAL: NCT02870816
Title: A Prospective, Randomized, Multi-Center Comparative Study of Amniotic Membrane Wound Graft Application Versus Tissue Engineered Skin Substitute in the Management of Non Healing Diabetic Foot Ulcers
Brief Title: Prospective, Comparitive, Randomized Study of Allograft Versus Skin Substitute in Non-healing Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professional Education and Research Institute (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTF-DFU-COMP-01
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tissue engineered skin substitute (Active Comparator): Application of tissue engineered skin substitute with Dressing Application, to be changed weekly following surgical debridement. Patient will practice Offloading. If the ulcer has not closed completely, an additional application of skin substitute will be applied weekly at weeks 2-11.
  Interventions: Procedure: Tissue Engineered Skin Substitute; Device: Offloading
- Amnionic membrane graft (Experimental): Application of amnionic membrane graft with Dressing Application, to be changed weekly following surgical debridement. Patient will practice Offloading. If the ulcer has not closed completely, an additional piece of amnionic membrane graft will be applied weekly at weeks 2-11
  Interventions: Device: Offloading; Procedure: Amnionic Membrane Graft

INTERVENTIONS:
Procedure: Tissue Engineered Skin Substitute — Application of skin substitute and non-adherent dressing, a moisture retentive dressing, and a multi-layer compression dressing.
  Arms: Tissue engineered skin substitute
Device: Offloading — Provision of offloading cast walker or similar sponsor-approved device. May convert into "instant total contact cast" and/or add felt/foam to supplement offloading.
Procedure: Amnionic Membrane Graft — Application of amnion membrane graft and non-adherent dressing, a moisture retentive dressing, and a multi-layer compression dressing.
  Arms: Amnionic membrane graft

SUMMARY:
The purpose of this study is to determine whether amnion membrane grafts are more effective than another tissue engineered skin substitute, when used to treat diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
Diabetes affects at least 9% of the population, or approximately 29 million people in the United States. Lower extremity ulcers are a serious complication for people with diabetes. Diabetic foot-related problems are the most frequent cause of hospitalization within this group and it is estimated that the total cost for treatment ranges from $10,000 to nearly $60,000 depending on ulcer severity and clinical outcomes. While many diabetic foot ulcers are superficial and can heal with conservative treatment, many are more severe and recalcitrant to standard of care (SOC). About a quarter of individuals with diabetes will develop a chronic non-healing ulcer over their lifetime and nearly 60 of every 10,000 individuals with diabetes will undergo a lower extremity amputation. Holzer and associates conducted a retrospective analysis of the costs for lower extremity ulcers in patients with diabetes and concluded that, given the high costs associated with treating these ulcers, the development of better treatment strategies is warranted. One such development in the treatment of chronic wounds is the use of amniotic membrane grafts. These materials have been used successfully for many years in the treatment of orthopedic, plastic/reconstructive, and urological applications. Initial studies have demonstrated the great success of amnionic membrane graft in the healing of chronic diabetic foot ulcers and it is believed that these grafts may be superior to older, more common skin substitutes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 or older
2. Informed consent must be obtained
3. Patient's ulcer must be diabetic in origin and larger than 1cm2. Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement.
4. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
5. Ulcer must be present for a minimum of four weeks duration, with documented failure of prior treatment to heal the wound.
6. Patient's ulcer must exhibit no clinical signs of infection.
7. Wound must be present anatomically on the foot as defined by beginning below the malleoli of the ankle
8. Additional wounds may be present but not within 3cm of the study wound
9. Patient is of legal consenting age.
10. Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
11. Serum Creatinine less then 3.0mg/dl.
12. HbA1c less than 12% taken prior to randomization .
13. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 90 days:

    1. Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
    2. ABIs with results of ≥0.7 and ≤1.2, OR
    3. Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg

Exclusion Criteria:

1. Patients presenting with an ulcer probing to bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients whose index diabetic foot ulcers are greater than 25cm2.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days.
4. Patients whose serum creatinine levels are 3.0mg/dl or greater as noted by serum blood testing within the last six months.
5. Patients with a known history of poor compliance with medical treatments.

6 Patients who are presently participating in another clinical trial.

7. Patients who are currently receiving radiation therapy or chemotherapy.

8. Patients with known or suspected local skin malignancy to the index diabetic ulcer.

9. Patients on anticoagulant medication will as in any surgical procedure, be monitored according to the protocols employed at the enrolling center.

10. Patients with uncontrolled autoimmune connective tissues diseases.

11. Non-revascularizable surgical sites.

12. Active infection at site.

13. Any pathology that would limit the blood supply and compromise healing.

14. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days.

15. Patient who are pregnant or breast feeding .

16. Patient who are taking medications that are considered immune system modulator.

17. Patient taking a cox-2 inhibitor.

18. Patient with wounds healing greater then 20% during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
The number of participants out of 60 with complete healing of their diabetic foot ulcers as measured by complete epithialization of the foot wound comparing the two active treatment groups | 6 weeks
  Examine the number of patient that go onto complete healing

SECONDARY OUTCOMES:
Number of wounds healed | 12 weeks
  examine the number of wounds that go on to complete healing
Time to healing/complete closure | 6 weeks
  examine the time it take for the patient to go onto complete healing
Time to healing/complete closure | 12 weeks
  examine the time it take for the patient to go onto complete healing
Cost effectiveness of each treatment modality. | 12 weeks
  Examine the cost to achieve closure in the wounds

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Chnari, PhD, Study Director — Director of Research and Development; Wound Care
Locations (3):
- United States (3):
  - Martinsville Research Institute, Martinsville, Virginia
  - Shenandoah Lower Extremity Research Institute, Roanoke, Virginia
  - Professional Education and Research Institute, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glat P, Orgill DP, Galiano R, Armstrong D, Serena T, DiDomenico LA, Kaufman J, Carter MJ, Jacobs AM, Zelen CM. Placental Membrane Provides Improved Healing Efficacy and Lower Cost Versus a Tissue-Engineered Human Skin in the Treatment of Diabetic Foot Ulcerations. Plast Reconstr Surg Glob Open. 2019 Aug 30;7(8):e2371. doi: 10.1097/GOX.0000000000002371. eCollection 2019 Aug. PMID 31592387
- See also: Publication of Clinical Study — https://journals.lww.com/prsgo/Fulltext/2019/08000/Placental_Membrane_Provides_Improved_Healing.20.aspx